CLINICAL TRIAL: NCT04996680
Title: Vascular Occlusion for Optimizing Functional Improvement in Patients With Knee Osteoarthritis
Acronym: VOFIKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-09925
Record Dates: First submitted 2021-07-12; First posted 2021-08-09 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Blood Flow Restriction
Keywords: Blood Flow Restriction; Strength training; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Assignment to the BFR or control group was stratified by sex (male/female/X) and affected leg (right, left, both), and only visible for physiotherapists treating patients. The study was single-blinded, as the outcome assessors were blinded from randomization whereas masking of participants was not possible due to the nature of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Blood flow restriction group (Experimental): patients in this group will undergo a standard strength training program combined with an occlusion cuff. The cuff will reduce the amount of blood flow and therefore increase the metabolic stimulus. The cuff will be used only during one quadriceps exercise, 2 times a week for 12 weeks.
  Interventions: Device: Blood Flow Restriction (by using smart-cuff pro devices, acting as pressurized tourniquet) combined low load strengh training
- Sham group (Sham Comparator): patients in this group will undergo the same standard strength training program as the BFR-group, combined with an occlusion cuff but pressurized so there is no significant effect on the lower limb blood flow. The cuff will be used only during one quadriceps exercise, 2 times a week for 12 weeks.
  Interventions: Device: Sham-BFR (by using smart-cuff pro devices, acting as pressurized tourniquet) combined with low load strength training
- Control group (Active Comparator): patients in this group will undergo the same standard strength training program as the BFR-group and placebo-group, but without a tourniquet.
  Interventions: Other: Standardised low load strength training

INTERVENTIONS:
Device: Blood Flow Restriction (by using smart-cuff pro devices, acting as pressurized tourniquet) combined low load strengh training — This group will undergo standard, traditional low load strength training consisting of calf, thigh, glute and core exercises, combined with optimal pressurized blood flow restriction
  Other Names: Kaatsu; partial vascular occlusion
  Arms: Blood flow restriction group
Other: Standardised low load strength training — This group will undergo standard, traditional low load strength training consisting of calf, thigh, glute and core exercises
  Arms: Control group
Device: Sham-BFR (by using smart-cuff pro devices, acting as pressurized tourniquet) combined with low load strength training — This group will undergo standard, traditional low load strength training consisting of calf, thigh, glute and core exercises, combined with blood flow restriction, but pressurized so the occlusion cuff has no significant effect on the lower limb blood flow.
  Arms: Sham group

SUMMARY:
Recent research in strength training physiology revealed that implementation of occlusion garments around the proximal aspect of the lower limbs in combination with low load strength training causes a reduced blood flow and thus providing a high metabolic stimulus, causing a training effect similar to high load training. This study will investigate the added effect of BFR focussing on functional outcome, pain-management and lower limb strength in patients with knee osteoarthritis. Therefore, 234 patiens will be divided into three equal groups (n=78), (control group, sham group and BFR-group) which will be subjected to a 12-week during standard strength training program, 2 times a week for 60 minutes. The first group, which will be submitted to low load resistance training commonly used in contemporary physiotherapy for OA, will serve as a control group whereas both the BFRT and Sham groups will objectify the additional value of implementing vascular occlusion in respective low load resistance training protocol.

DETAILED DESCRIPTION:
Recent research in strength training physiology, revealed that implementation of occlusion garments around the proximal aspect of the segment submitted to strength training (i.e. the upper thigh, in case of lower limb and knee joint training) results in significant increments in metabolic and mechanical muscle loading, facilitating neuromuscular responses in terms of muscle fiber recruitment and muscle fiber hypertrophy/gains in muscle mass, even at fairly low training dosages (<50% of 1RM). As a consequence, BFR guided resistance training at low training intensities renders a training response similar to what can be expected from high intensity strength training. Occlusion at the proximal site of the segment submitted to strength training, reduces both vascular in- and outflow. This reduced blood flow is thought to induce an ischemic/hypoxic environment that enhances the training effect in the exercising muscle, leading to increased muscle mass and strength. In accordance with this theoretic framework, results of a recent study which compared the training effects between High Intensity Resistance Training (HIRT), Low Intensity Resistance Training (LIRT) and Low Intensity Resistance Training with BFR (BFRT), demonstrated that both the HIRT and the BFRT resulted in similar significant improvements in 1RM knee extension strength, functional performance and Quadriceps Cross Sectional Area (CSA), whereas no differences were found after a 12 week period of LIRT. On the contrary, pain scores objectified by means of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) significantly reduced in the BFRT, whereas this was not the case for the HIRT group in which 4 patients were also excluded due to the onset of exercise-induced knee pain. Although previous scientific research has already provided a quite solid proof of concept by assessing the short term results of BFR training in small sample sizes of patients at risk of or suffering from knee OA, ready-to-use guidelines and specific implementation instructions of BFR-based physical therapy and strength training are non-existent at present. With this TBM project, it is our intention to reinforce the scientific evidence regarding the substantial benefits and significant added value of BFR-guided low intensity resistance training in both the stabilization and rehabilitation of knee osteoarthritis, as well as to provide the clinicians ((para)medics and trainers) in hospital, clinical practice and fitness/training settings with specific guidelines with regard to practical implementation of respective exercise protocols.

This will be done using a large scale Randomized Clinical Trial Design in which a standardized strength training protocol will be implemented for functional rehabilitation purposes in a population of 234 participants diagnosed with knee OA, using three different loading categories:

* (n=78) Low Load Resistance Training (Control)
* (n=78) Blood Flow Restricted Low Load Resistance Training (BFRT)
* (n=78) Low Load Resistance Training with sham BFR component (Sham). The first group, which will be submitted to low load resistance training commonly used in contemporary physiotherapy for OA, will serve as a control group whereas both the BFRT and Sham groups will objectify the additional value of implementing vascular occlusion in respective low load resistance training protocol.

The intervention consists of a 12 week during standardised strength program, 2 times a week for 60 minutes. To evaluate and objectify any training effect, patient overall Quality of Life (QoL) and knee function, 4 screening moments are planned; at baseline (week 0), after 6 weeks, post intervention (13 weeks) and a follow-up screening after 6 months to assess the retention effect and thus, the sustainability of this training modality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee osteoarthritis
* Speak Dutch, French or English
* No other pathology restricting patients to participate safe
* Time and motivation to visit 2x/w for 12 weeks

Exclusion Criteria:

* Neurological disorders
* previous surgery or disorder with blood vessels.
* (Symptomatic) heart or vascular disease
* Increased risk for DVT
* Avoiding physical exercise due to medical conditions.
* Rheumatoid arthritis
* BMI >30
* Recent severe trauma or surgery in the lower extremity

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Assessing change within Knee Injury and Osteoarthritis Outcome Score (KOOS) | assessing change at 4 time points; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  A comprehensive analysis of patient function at level of activities of daily living as well as in sports participation. KOOS consists of 5 subscales: (1) Pain, (2) other Symptoms, (3) Function in daily living (ADL), (4) Function in sport and recreation (Sport/Rec) and (5) knee related Quality of life (QOL).

SECONDARY OUTCOMES:
Assessing change within Pain Catastrophizing Scale (PCS) | 4 times; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  The Pain Catastrophizing Scale (PCS) will evaluate the patient's tendency towards pain catastrophizing and risk of developing chronic pain, and as such the quality of the patients psychosocial health status.
Assessing change within thigh muscle strength | assessing change at 4 time points; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  objectified by means of Hand Held Dynamometry (HHD) assessment (maximal isometric muscle strength) of the quadriceps and hamstring muscle. Each muscle will be tested in a standardized fashion and sequence. The patient will be informed about the purpose and the content of each strength test, after which the investigator will demonstrate which muscle will be tested, the starting position that should be adopted as well as the specific location and direction at/in which the static resistance will be applied. Afterwards, the participants will be tested once at submaximal and twice at maximal level of isometric strength output, after which the best trial will be taken into account for data registration and processing.
Assessing change within Single leg Hop for Distance (SHD) | assessing change at 4 time points; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  unilateral jump and landing. Patient get 3 attempts on both sides
Assessing change within Knee Bent Test (KBT) | assessing change at 4 time points; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  unilateral knee flexion and extension (~unilateral squat)
Assessing change within 6 minute walk test (6MWT) | assessing change at 4 time points; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  walk as far as possible within 6 minutes. Patient is allowed to take a break during the test, although time keeps counting down.
Assessing change within 40m FPWT | assessing change at 4 time points; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  40m walking as fast as possible
Assessing change within chair stand test | assessing change at 4 time points; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  go from sit (on a chair) to stand as much as possible within 30 seconds
assessing change within stair climb test | assessing change at 4 time points; 1) baseline screening (week 0), 2) after 6 weeks, 3) post intervention after 13 weeks and 4) follow-up screening after 24 weeks.
  go 11 steps upwards and downwards on a stair as fast as possible (although safe)
Assessing change within International physical activity questionnaire (IPAQ) | assessing change every week, starting from baseline (Week 0) until the follow-up after 24 weeks.
  The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity from the last 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Erik Witvrouw, Prof. dr., Study Chair — Rehabilitation science & Physiotherapy Ghent University; Jan Victor, Prof. Dr., Principal Investigator — Orthopedics & Traumatology Ghent University Hospital
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

REFERENCES:
- [Derived] Jacobs E, Stroobant L, Witvrouw E, Victor J, Acx F, van der Jeugt J, Schuermans J, Wezenbeek E. Sustained benefits of blood flow restriction therapy in knee osteoarthritis rehabilitation: 1-year follow-up of a randomised controlled trial. Br J Sports Med. 2025 Nov 26;59(21):1481-1489. doi: 10.1136/bjsports-2024-109524. PMID 40846463
- [Derived] Jacobs E, Stroobant L, Victor J, Elewaut D, Tampere T, Wallaert S, Witvrouw E, Schuermans J, Wezenbeek E. Vascular occlusion for optimising the functional improvement in patients with knee osteoarthritis: a randomised controlled trial. Ann Rheum Dis. 2025 Feb;84(2):341-350. doi: 10.1136/ard-2024-226579. Epub 2025 Jan 2. PMID 39919906
- [Derived] Jacobs E, Rolnick N, Wezenbeek E, Stroobant L, Capelleman R, Arnout N, Witvrouw E, Schuermans J. Investigating the autoregulation of applied blood flow restriction training pressures in healthy, physically active adults: an intervention study evaluating acute training responses and safety. Br J Sports Med. 2023 Jul;57(14):914-920. doi: 10.1136/bjsports-2022-106069. Epub 2023 Jan 5. PMID 36604156